CLINICAL TRIAL: NCT06939140
Title: Predictors of Urinary Incontinence After Endoscopic Transurethral Bipolar Prostatectomy: a Prospective Cohort Study
Brief Title: Urinary Incontinence After Endoscopic Prostatectomy
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mostafa Mohamed Atef Abdelaziz Mostafa, Lecturer of Urology, Assiut University
Other Study IDs: UI after prostatectomy
Record Dates: First submitted 2025-04-15; First posted 2025-04-22 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Urinary Incontinence (UI)
Keywords: Stress Urinary Incontinence (SUI); Urge Urinary Incontinence (UUI); Benign Prostatic Hyperplasia (BPH); Bipolar enucleation of the Prostate (BipolEP); Bipolar transurethral reaction of the prostate (B-TURP)
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress; Urinary Incontinence, Urge; Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic transurethral bipolar prostatectomy patients: Benign Prostatic Hyperplasia patients who will undergo endoscopic transurethral bipolar prostatectomy
  Interventions: Procedure: Bipolar prostatectomy

INTERVENTIONS:
Procedure: Bipolar prostatectomy — Endoscopic transurethral bipolar enucleation or reaction of the prostate

SUMMARY:
This is a prospective cohort study aiming to identify the preoperative and intraoperative predictors of urinary incontinence after endoscopic transurethral bipolar prostatectomy

DETAILED DESCRIPTION:
Benign prostatic hyperplasia (BPH) represents a progressive, age-related proliferation of prostatic stromal and epithelial cells, with histopathological changes typically manifesting after the fourth decade of life. Epidemiological studies demonstrate a prevalence increasing from approximately 50% in men aged 60 years to 90% by age 85 years. The condition frequently results in bladder outlet obstruction, clinically presenting as lower urinary tract symptoms (LUTS) that are conventionally categorized into obstructive (voiding) and storage (irritative) subtypes. Among contemporary surgical interventions, transurethral bipolar prostatectomy techniques - including bipolar transurethral resection of the prostate (B-TURP) and bipolar laser enucleation of the prostate (BipoLEP) - have established efficacy in the management of BPH-induced LUTS, as demonstrated in randomized controlled trials and meta-analyses.

Postoperative urinary incontinence (UI) remains among the most clinically significant complications following surgical management of benign prostatic hyperplasia (BPH). Early transient UI represents a frequently observed postoperative sequela, serving as both a primary source of patient anxiety regarding surgical intervention and a substantial determinant of postoperative dissatisfaction. While the majority of transient UI cases demonstrate spontaneous resolution within 1-6 months postoperatively, persistent UI develops in a clinically relevant subset of patients. This chronic manifestation constitutes a serious long-term complication which decrease the quality of life of the patients.

Reported rates of urinary incontinence following BPH surgery exhibit considerable variability, which may be attributed to differences in surgical techniques, inconsistent definitions of incontinence, and heterogeneity in assessment methods. Moreover, the majority of studies fail to specify the type or duration of incontinence.

Predictors of postoperative urinary incontinence (UI) following endoscopic surgery for BPH require systematic evaluation to optimize preoperative counseling and identify high-risk patients. A thorough discussion of UI risk should be incorporated into the shared decision-making process. This prospective study aims to identify and characterize preoperative and intraoperative risk factors for stress (SUI) and urge (UUI) urinary incontinence in patients undergoing endoscopic BPH surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Males ≥50 years undergoing primary B-TURP/BipolEP for BPH
* Preoperative IPSS ≥8, Qmax ≤15 mL/s, prostate volume ≥30mL
* No prior incontinence/neurological bladder dysfunction

Exclusion Criteria:

* Prostate cancer history
* Concurrent anti-incontinence procedures

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Benign prostatic hyperplasia patients who will undergo endoscopic bipolar transurethral prostatectomy and develop urinary incontinence will be included in the study. Their preoperative and intraoperative data will be studied to identify if there is association between their preoperative and intraoperative parameters and the development of urinary incontinence after endoscopic bipolar transurethral prostatectomy
Sampling Method: Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Preoperative predictors of urinary incontinence | At 6 months after the procedure
  Association between patients' preoperative parameters and occurrence of urinary incontinence after the procedure

SECONDARY OUTCOMES:
Intraoperative predictors of urinary incontinence | At 6 months after the procedure
  Association between intraoperative parameters and occurrence of urinary incontinence after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Urology Hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be made available to protect privacy of patients

REFERENCES:
- [Background] Matsushita K, Kent MT, Vickers AJ, von Bodman C, Bernstein M, Touijer KA, Coleman JA, Laudone VT, Scardino PT, Eastham JA, Akin O, Sandhu JS. Preoperative predictive model of recovery of urinary continence after radical prostatectomy. BJU Int. 2015 Oct;116(4):577-83. doi: 10.1111/bju.13087. Epub 2015 Mar 30. PMID 25682782
- [Background] Castellani D, Rubilotta E, Fabiani A, Maggi M, Wroclawski ML, Teoh JY, Pirola GM, Gubbiotti M, Pavia MP, Gomez-Sancha F, Galosi AB, Gauhar V. Correlation Between Transurethral Interventions and Their Influence on Type and Duration of Postoperative Urinary Incontinence: Results from a Systematic Review and Meta-Analysis of Comparative Studies. J Endourol. 2022 Oct;36(10):1331-1347. doi: 10.1089/end.2022.0222. Epub 2022 Jun 13. PMID 35587146
- [Background] Bauer RM, Gozzi C, Hubner W, Nitti VW, Novara G, Peterson A, Sandhu JS, Stief CG. Contemporary management of postprostatectomy incontinence. Eur Urol. 2011 Jun;59(6):985-96. doi: 10.1016/j.eururo.2011.03.020. Epub 2011 Mar 21. PMID 21458914
- [Background] Sandhu JS, Breyer B, Comiter C, Eastham JA, Gomez C, Kirages DJ, Kittle C, Lucioni A, Nitti VW, Stoffel JT, Westney OL, Murad MH, McCammon K. Incontinence after Prostate Treatment: AUA/SUFU Guideline. J Urol. 2019 Aug;202(2):369-378. doi: 10.1097/JU.0000000000000314. Epub 2019 Jul 8. PMID 31059663
- [Background] Huang X, Chen XX, Chen X, Chen QZ, Wang L, Li C, Tian JL. Feasibility of anterior lobe-preserving transurethral enucleation and resection of prostate on improving urinary incontinence in patients with benign prostatic hyperplasia: A retrospective cohort study. Medicine (Baltimore). 2023 Feb 17;102(7):e32884. doi: 10.1097/MD.0000000000032884. PMID 36800610
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Background] Magistro G, Schott M, Keller P, Tamalunas A, Atzler M, Stief CG, Westhofen T. Enucleation vs. Resection: A Matched-pair Analysis of TURP, HoLEP and Bipolar TUEP in Medium-sized Prostates. Urology. 2021 Aug;154:221-226. doi: 10.1016/j.urology.2021.04.004. Epub 2021 Apr 21. PMID 33891930
- [Background] Pagano E, Laudato M, Griffo M, Capasso R. Phytotherapy of benign prostatic hyperplasia. A minireview. Phytother Res. 2014 Jul;28(7):949-55. doi: 10.1002/ptr.5084. PMID 25165780